CLINICAL TRIAL: NCT02935998
Title: A Multi-Center,Open-Labeled,Intervention Study:The Efficacy And Safety Of Intramuscular Ziprasidone For Three Days In Patients With Psychotic Agitation
Brief Title: The Efficacy And Safety Of Intramuscular Ziprasidone For Three Days In Patients With Psychotic Agitation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yang Fude (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor-Investigator, Yang Fude, A Multi-Center,Open-Labeled,Intervention Study:The Efficacy And Safety Of Intramuscular Ziprasidone For Three Days In Patients With Psychotic Agitation, Beijing HuiLongGuan Hospital
Organization: Beijing HuiLongGuan Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QLXTJY-201649
Record Dates: First submitted 2016-10-14; First posted 2016-10-18 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-09

CONDITIONS: Schizophrenia
Keywords: schizophrenia; agitation; ziprasidone
MeSH Terms: conditions — Schizophrenia; Psychomotor Agitation | interventions — ziprasidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ziprasidone (Experimental): The injection mesylate ziprasidone used in this study have been marketed, manufactured by Pfizer and provided study drug for research purposes.Strength:Each vial contains Ziprasidone 30 mg, Sulfobutyl betadex sodium 441 mg. When reconstituted as directed the solution for injection contains the equivalent of 20 mg per mL of Ziprasidone.The initial dosage of ziprasidone injection：Most patients are suggested with 20mg i.m. Those with first-episode, lower age, emaciated body, or BARS score at 5 are suggest with 10mg i.m. Doses of 10 mg may be administered every two hours; doses of 20 mg may be administered every four hours up to a maximum of 40 mg/day.
  Interventions: Drug: Ziprasidone

INTERVENTIONS:
Drug: Ziprasidone — During the study, at least 1 injection is needed per day. Whether the second, third or fourth one is needed according to patients' symptoms. If the BARS score>=5, clinicians are supposed to give 10mg or 20mg.If lower than 5, clinicians could choose to give 10mg or not according to patients' symptoms and doctor's experience. Doses of 10 mg may be administered every two hours; doses of 20 mg may be administered every four hours up to a maximum of 40 mg/day.It is not recommended to combine with other oral antipsychotic drugs. But if the patients' daily dose of injection has reached 40mg and agitation occurred 4 hours later after the last injection, with the BARS score higher than 5.The clinicians can determine whether or not to combine oral antipsychotic drug, and the dosage.
  Other Names: Injection mesylate ziprasidone

SUMMARY:
1. The title of this study is a multi-center,non randomized,open-labeled,intervention study:the efficacy and safety of intramuscular ziprasidone for three days in patients with acute psychotic agitation.
2. The primary objectiveis to evaluate the efficacy of intramuscular ziprasidone in patients with acute psychotic agitation in daily clinical practice.
3. The secondary objectives are:1.To evaluate the safety of intramuscular ziprasidone in patients with acute psychotic agitation in daily clinical practice.2.To compare the efficacy and tolerance of intramuscular ziprasidone in patients with agitation in the different psychotic disorder 3.To compare the efficacy and tolerance of intramuscular ziprasidone in patients with first episode andmulti-episode patients. 4.To explore the measured based administration according to severity of symptoms.5.To compare the efficacy and tolerance of ziprasidone im between the monotherapy and combination with other antipsychotic drug in clinical practice.
4. The Rationale:In China, the studies of ziprasidone im treating agitation focus on schizophrenia. But in the foreign country, ziprasidone im also is approved to treat psychotic agitation, including bipolar and schizoaffective disorder. And in the clinical practice of China, ziprasidone im is also used to treat other patients, although the evidence is less. In this study, we assume ziprasidone im treat the psychotic agitation is effective and safe.
5. Study populations:The study plan to enroll 1000 subjects in China. （6）The background and the hypothesis：The researches of ziprasidone mesylate injection in our country are more concentrated in schizophrenia at present, while in foreign countries ziprasidone is approved for psychotic agitation, including mania etc. It's also used for substance abuse and alcohol induced agitation.Therefore, this study assumes that ziprasidone mesylate injection is effective in the treatment of acute agitation, and it's well tolerated.

DETAILED DESCRIPTION:
1. Trial Design:This is a multi-center, open-labeled, intervention study.
2. STUDY EVALUATION：1)Primary efficacy endpoint：The change of BARS total scores from baseline to the endpoint.2)Secondary efficacy endpoint：

   * The change of CGI-S from baseline to the endpoint
   * The change of BARS/CGI-S/CGI-I from baseline to every visit
   * The percentage of response at the end of 2h(BARS decreased score>=2)
   * Subgroup analysis:(1)Comparison of the difference of the reduction in BARS/CGI-S in the different diseases subgroup.(2)Comparison of the difference of the reduction in BARS/CGI-S in the first episode and multi-episode patients.(3)Comparison of the difference of the reduction in BARS/CGI-S in the different previous antipsychotic treatment.(4)Comparison of the difference of disease categories, dosage, duration, and the reduction in BARS/CGI-S in the monotherapy and combination with other oral antipsychotic drugs Safety evaluation 3)Include adverse events, ECG(the change rate of ECG and the average change of QT),vital signs from the baseline to the endpoint.

     1. The change of Simpson-Angus with from the baseline to endpoint.
     2. The incidence of ADR、extrapyramidal symptoms、tachycardia during the studyThe incidence of during the study.
3. STUDY DRUGS:The injection mesylate ziprasidone used in this study have been marketed, manufactured by Pfizer and provided study drug for research purposes.Strength:Each vial contains Ziprasidone 30 mg, Sulfobutyl betadex sodium 441 mg. When reconstituted as directed the solution for injection contains the equivalent of 20 mg per mL of Ziprasidone.Ziprasidone intramuscular is intended for intramuscular use only and should not be administered intravenously.
4. DATA ADMINISTRATION AND STATISTICAL METHODS:The case report form (CRF) used in this clinical study is in paper form.

   The data and statistical analysis collected in study will be recorded in the statistical analysis program (SAP).
5. Basic principles of research design:Collecting the safety, effectiveness indexes in the process of drug treatment, analysis the changes before and after 3 days of the treatment, and record injection in the process of the study, in order to analyze the safety and efficacy of injection ziprasidone in the real clinical practice.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet the following criteria to be enrolled in the study:

* Male or female subjects aged 18-65 years
* Inpatients and outpatients who meet the diagnostic criteria for schizophrenia, schizoaffective disorder, Bipolar disorder with manic features or mixed features according to ICD-10
* BARS score >= 5 at baseline；
* Female subjects must have effective means of contraception (for example, oral prescription contraceptives, contraceptives, intrauterine device, a male partner sterilization, etc.) before screening phase and during the whole duration of study;
* Subjects can comply with the visit plan, treatment, laboratory examination and other research program;
* Subjects or their legal representatives understand the content of this research, agreed to participate in and sign a written informed consent and dated.

Exclusion Criteria:

* Subjects who meet any of the following criteria will be excluded from the study:
* Have any major or unstable cardiovascular (especially arrhythmia), respiratory, nervous system, including epilepsy or obvious cerebrovascular disease), kidney, liver, endocrine, immune disease or related illness
* Have myocardial infarction or decompensated heart failure recently
* Confirmed clinically significant abnormal laboratory values
* Clinically significant ECG abnormality
* Subjects with a history of QTc prolongation or a pre-drug QTc of 450 msec or greater
* Subjects with serum K+ or Mg2+ out of the normal range
* A history of malignant syndrome or tardive dyskinesia history
* Concomitant use of drugs which may induce QTc prolongation during the study ,such as Sotalol, quinidine, amiodarone, erythromycin, clozapine and clomipramine
* Known allergy to ziprasidone or any product ingredient
* Pregnant or lactating women or decide to pregnant in 3 month
* Use of antipsychotic agents within 12 hours or parenteral benzodiazepines within 4 hours prior to the baseline.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
The change of BARS total scores | 3 days after the first shot

SECONDARY OUTCOMES:
The change of CGI-S scores | 3 days after the first shot

OTHER OUTCOMES:
The change of BARS/CGI-S/CGI-I scores from baseline to every visit | 3 days after the first shot
The percentage of response at the end of 2h(BARS decreased score>=2) | 2 hours after the first shot
The change of Simpson-Angus scores with from the baseline to endpoint | 3 days after the first shot
The incidence of ADR during the study in percent | 3 days after the first shot
The incidence of extrapyramidal symptoms during the study in percent | 3 days after the first shot
The incidence of tachycardia during the study in percent | 3 days after the first shot
The significance change rate of ECG and the average change of QT | 3 days after the first shot

CONTACTS AND LOCATIONS:
Overall Officials: Yang Fude, director, Principal Investigator — Beijing HuiLongGuan Hospital
Locations (1):
- Beijing Huilongguan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Marder SR. A review of agitation in mental illness: treatment guidelines and current therapies. J Clin Psychiatry. 2006;67 Suppl 10:13-21. PMID 16965191
- [Result] Zhang H, Wang G, Zhao J, Xie S, Xu X, Shi J, Deng H, Li K, Gao C, Wang X, Vanderburg D, Pan S, Tang H, Shu L, Karayal ON. Intramuscular ziprasidone versus haloperidol for managing agitation in Chinese patients with schizophrenia. J Clin Psychopharmacol. 2013 Apr;33(2):178-85. doi: 10.1097/JCP.0b013e3182839612. PMID 23422376
- [Result] Zimbroff DL, Allen MH, Battaglia J, Citrome L, Fishkind A, Francis A, Herr DL, Hughes D, Martel M, Preval H, Ross R. Best clinical practice with ziprasidone IM: update after 2 years of experience. CNS Spectr. 2005 Sep;10(9):1-15. doi: 10.1017/s1092852900025487. PMID 16247923